CLINICAL TRIAL: NCT03104842
Title: Clinical Phase II, Multicenter, Open-label Study Evaluating iNduction, Consolidation and Maintenance With Isatuximab (SAR650984), Carfilzomib, LEnalidomide and Dexamethasone (I-KRd) in Primary Diagnosed High-risk Multiple Myeloma paTients
Brief Title: Evaluation iNduction, Consolidation and Maintenance Treatment With Isatuximab , Carfilzomib, LEnalidomide and Dexamethasone
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG-CONCEPT
Record Dates: First submitted 2017-03-29; First posted 2017-04-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Cytogenetic High-Risk
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Transplantation (Experimental): Patients ≤ 70 years of age and eligible for stem cell transplantation will enter study arm A They will undergo 6 cycles of Induction Treatment : Carfilzomib, Lenalidomid, Isatuximab (I-KRd), after intensification another 4 cycles of I-KRd as consolidation will be followed by IKR maintenance until PD or Toxicity
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- Arm B No-Transplantation (Experimental): Patients > 70 years or ineligible for stem cell transplantation will enter study arm B They will undergo 12 cycles of Treatment : Carfilzomib, Lenalidomid, Isatuximab (I-KRd) (6 Cycles Induction, 2 Cycles Intensification, 4 Cycles Consolidation),to be followed by I-KR maintenance util PD or Toxicity
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Antibody Intravenous
Drug: Carfilzomib — Intravenous
Drug: Lenalidomide — Capsel
Drug: Dexamethasone — Capsel

SUMMARY:
A Clinical Phase II, multicenter, Open-label study evaluating iNduction, consolidation and maintenance treatment with Isatuximab (SAR650984), Carfilzomib, LEnalidomide and Dexamethasone (I-KRd) in Primary diagnosed high-risk multiple myeloma paTients

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have newly diagnosed, untreated, symptomatic (according to the revised CRAB criteria 2014), documented myeloma and have measurable disease (serum M-protein ≥ 1 g/dL (for IgA ≥ 0.5 g/dL) or urine M-protein ≥ 200 mg/24 hours) or in case of oligosecretory myeloma: involved FLC level ≥ 10 mg/dl, provided sFLC ratio is abnormal or in case of asecretory myeloma: > 1 focal lesions measurable by MRI

   Subjects must have high-risk myeloma defined as followed:
   * Presence of one or more of the following cytogenetic abnormalities (determined by FISH):

     * Del(17p) in ≥ 10% of purified cells
     * t(4;14)
     * ≥ 3 copies +1q21
     * t(14;16)
   * ISS Stage II or III (all patients)
   * FISH analysis of external laboratories other than Heidelberg is accepted, a list of laboratories will be filed in the study central.
2. Must be ≥ 18 years at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements in the investigators opinion.
4. WHO performance status 0-3 (WHO=3 is allowed only if caused by MM and not by co-morbid conditions)
5. Females of childbearing potential (FCBP) (1) must agree to refrain from becoming pregnant for 28 days prior to initiation of study drug, while on study drug and for 150 days* after discontinuation from the study drug by using 2 reliable methods of contraception and must agree to regular pregnancy testing during this timeframe.

   * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months) 3) has achieved menarche at some point.
6. Females must agree to abstain from breastfeeding during study participation and 30 days* after study drug discontinuation.
7. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 150 days* following discontinuation from this study, even if he has undergone a successful vasectomy.
8. Males must also agree to refrain from donating semen or sperm while on treatment with any study drug and for 150 days* after discontinuation from this study treatment.
9. All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
10. All subjects must agree not to share medication.
11. All participating subjects have to follow the requirements of the Lenalidomide Pregnancy Prevention Plan

Exclusion Criteria:

1. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize Carfilzomib), mannitol, sucrose, histidine (as base and hydrochloride salt) and polysorbate 80 or any of the components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
2. Patients with known systemic amyloidosis (except for AL amyloidosis of the skin or the bone marrow)
3. Administration of systemic chemotherapy, biological, immunotherapy or any investigational agent (therapeutic or diagnostic) for multiple myeloma except bisphosphonate therapy. Emergency treatment with dexamethasone is allowed when the cumulative dexamethasone dose is less or equal 160 mg. It is allowed to include patients in the trial after 1 cycle (4 weeks) of any anti-myeloma first-line treatment.
4. Any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,000/μL, unless related to myeloma
   * Platelet count < 30,000/ μL (in case of platelets < 50.000 /µl and ≥ 30.000 /µl myeloma bone marrow infiltration should be ≥ 50%)
   * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L); or free ionized calcium > 6.5 mg/dL (> 1.6 mmol/L)
   * Serum GOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN) or serum total bilirubin > 2.0 mg/dL if not due to hereditary abnormalities as Gilbert's disease or hereditary hemolysis (Note: if the mentioned limits for bilirubin or ASAT/ALAT are exceeded, but there is no significant hepatic dysfunction at investigator's discretion, the study office has to be consulted prior to inclusion)
   * Patients with severe renal impairment (eGFR < 30 ml/min/1.73 m², MDRD formula or CDK-EPI or Creatinine Clearance < 30 ml/min)
5. Active congestive heart failure (NYHA Class III to IV), symptomatic cardiac ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within four months prior study entry.
6. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B sAg and core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed).
7. Acute active, uncontrolled infection
8. Significant neuropathy (Grades 3 to 4, or Grade 2 with pain according CTC V4.03)
9. Second malignancy within the past 5 years except:

   * adequately treated basal cell or squamous cell skin cancer
   * carcinoma in situ of the cervix
   * prostate cancer Gleason Score ≤ 6 with stable PSA over the past 12 months
   * breast carcinoma in situ with full surgical resection
   * treated medullary or papillary thyroid cancer
10. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to study entry.
11. Major surgery within 4 weeks prior to cycle 1 day 1 (kyphoplasty is not considered major surgery); subjects should have been fully recovered from any surgical related toxicities.
12. Female patients who are pregnant or lactating
13. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.
14. Participation in any other clinical trial (with the exclusion of observational, non-interventional studies))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
MRD negativity | after consolidation , an average of 1 year from first dosis
  MRD negativity (8-color flow, Euro-Flow plus Black Swan Panel)

CONTACTS AND LOCATIONS:
Overall Officials: Katja Weisel, Prof, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (17):
- Germany (17):
  - Vivantes Am Urban, Berlin
  - Campus Benjamin Franklin Charite Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Städt. Kliniken Bielefeld Klinikum Mitte, Bielefeld
  - Johanniter-Krankenhaus Bonn, Bonn
  - Uniklinikum Chemnitz, Chemnitz
  - Uniklinik Köln, Cologne
  - St. Antonius Hospital, Eschweiler
  - Universitätsklinikum Essen, Essen
  - Asklepios Altona, Hamburg
  - University Hospital Hamburg Eppendorf, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Philipps-Universität Marburg, Marburg
  - Kliniken Maria Hilf GmbH, Klinik für Hämatologie, Onkologie und Gastroenterologie, Mönchengladbach
  - Klinikum Osnabrück, Osnabrück
  - Universitätsklinikum Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leypoldt LB, Besemer B, Asemissen AM, Hanel M, Blau IW, Gorner M, Ko YD, Reinhardt HC, Staib P, Mann C, Lutz R, Munder M, Graeven U, Peceny R, Salwender H, Jauch A, Zago M, Benner A, Tichy D, Bokemeyer C, Goldschmidt H, Weisel KC. Isatuximab, carfilzomib, lenalidomide, and dexamethasone (Isa-KRd) in front-line treatment of high-risk multiple myeloma: interim analysis of the GMMG-CONCEPT trial. Leukemia. 2022 Mar;36(3):885-888. doi: 10.1038/s41375-021-01431-x. Epub 2021 Nov 3. No abstract available. PMID 34732857
- [Result] Leypoldt LB, Tichy D, Besemer B, Hanel M, Raab MS, Mann C, Munder M, Reinhardt HC, Nogai A, Gorner M, Ko YD, de Wit M, Salwender H, Scheid C, Graeven U, Peceny R, Staib P, Dieing A, Einsele H, Jauch A, Hundemer M, Zago M, Pozek E, Benner A, Bokemeyer C, Goldschmidt H, Weisel KC. Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone for the Treatment of High-Risk Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2024 Jan 1;42(1):26-37. doi: 10.1200/JCO.23.01696. Epub 2023 Sep 27. PMID 37753960
- [Derived] Leypoldt LB, Tichy D, Besemer B, Hanel M, Raab MS, Mann C, Munder M, Reinhardt HC, Nogai A, Gorner M, Ko YD, de Wit M, Salwender H, Scheid C, Graeven U, Peceny R, Staib P, Dieing A, Einsele H, Jauch A, Hundemer M, Zago M, Pozek E, Benner A, Bokemeyer C, Goldschmidt H, Weisel KC. Plain language summary of isatuximab plus carfilzomib, lenalidomide, and dexamethasone for the treatment of people with high-risk newly diagnosed multiple myeloma. Future Oncol. 2024 Dec;20(39):3193-3207. doi: 10.1080/14796694.2024.2402639. Epub 2024 Sep 30. PMID 39345094
- [Derived] Oliva S, Kaiser MF. Is it time to tailor treatment on the basis of minimal residual disease in multiple myeloma? Lancet Haematol. 2021 Dec;8(12):e876-e877. doi: 10.1016/S2352-3026(21)00341-0. No abstract available. PMID 34826409
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481